CLINICAL TRIAL: NCT02575755
Title: A Safety, Tolerability, Pharmacokinetic and Efficacy Study of Azithromycin Plus Piperaquine as Presumptive Treatment in Pregnant Papua New Guinean Women
Brief Title: A Safety, Tolerability, Pharmacokinetic and Efficacy Study of Azithromycin Plus Piperaquine as Presumptive Treatment in Pregnant PNG Women
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Papua New Guinea Institute of Medical Research (Other Government)
Collaborators: The University of Western Australia (Other); University of Melbourne (Other); Malaria in Pregnancy Consortium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MRAC10.53
Record Dates: First submitted 2015-10-08; First posted 2015-10-15 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Pregnancy; Infections, Plasmodia; Drug Kinetics; Clinical Efficacy
Keywords: Azithromycin; Piperaquine; IPTp; Pharmacokinetics; Efficacy
MeSH Terms: conditions — Infections | interventions — Azithromycin; piperaquine; fanasil, pyrimethamine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Efficacy Study: Azithromycin plus piperaquine (Experimental): At baseline, participants receive three daily doses (0, 24 and 48 hours) of i) 1 g azithromycin as 2 x film-coated 500 mg tablets ii) 960 mg piperaquine tetraphosphate tablets as 3 x 320 mg tablets
  Interventions: Drug: Azithromycin plus piperaquine phosphate
- Efficacy Study Control: National Standard Treatment (Active Comparator): At baseline, participants receive a single dose of sulfadoxine-pyrimethamine comprising 1,500 mg of sulfadoxine and 75 mg pyrimethamine in tablet form
  Interventions: Drug: Sulfadoxine-pyrimethamine
- Pharmacokinetic Study: Azithromycin plus piperaquine (Experimental): At baseline, participants receive three daily doses (0, 24 and 48 hours) of i) 1 g azithromycin as 2 x film-coated 500 mg tablets ii) 960 mg piperaquine tetraphosphate tablets as 3 x 320 mg tablets
  Interventions: Drug: Azithromycin plus piperaquine phosphate

INTERVENTIONS:
Drug: Azithromycin plus piperaquine phosphate
  Other Names: Sandoz Azithromycin; Sigma-Tau Piperaquine tetraphosphate
  Arms: Efficacy Study: Azithromycin plus piperaquine; Pharmacokinetic Study: Azithromycin plus piperaquine
Drug: Sulfadoxine-pyrimethamine
  Arms: Efficacy Study Control: National Standard Treatment

SUMMARY:
Plasmodium falciparum parasitaemia in pregnancy is associated with maternal anaemia, low birth-weight and increased perinatal mortality. Whilst continuous prophylaxis is difficult to implement, intermittent presumptive treatment in pregnancy (IPTp) has proved to be practical and effective. In PNG, pregnant women currently receive IPTp using sulfadoxine-pyrimethamine, however, this therapy has the potential to be compromised by parasite resistance.

The aim of the present trial is to assess the safety, tolerability, pharmacokinetics and efficacy of azithromycin (AZI) plus piperaquine (PQ) given as IPTp to pregnant Papua New Guinea women. The study will comprise of two sub-studies:

(i) A safety, tolerability and pharmacokinetic study of AZI-PQ in pregnancy. (ii) A safety, tolerability and preliminary efficacy study of AZI-PQ in pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* >14 weeks and <30 weeks gestation
* No signs of severe malaria by World Health Organisation criteria
* No significant concomitant disease (such as TB)
* No prior history of an adverse reaction to AZI or PQP
* No prior treatment with these drugs in the past 4 weeks
* Can attend all follow-up visits
* Provide informed consent

Exclusion Criteria:

* Have signs of severe malaria by WHO criteria
* Significant concomitant disease such as TB as assessed by the attending clinician
* A history/family history of sudden death or of congenital prolongation of the QTc interval
* Any clinical condition known to prolong the QTc interval
* A history of complicated pregnancies/deliveries
* A prior history of an adverse reaction to AZI or PQP
* Have taken these drugs in the past 4 weeks
* Cannot attend any of the follow-up visits
* Do not provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-10; Primary Completion 2016-07 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Efficacy of azithromycin plus piperaquine for the prevention of malaria during pregnancy | 42 days intensive follow-up, final end-point at 2 weeks post delivery
  The efficacy of azithromycin plus piperaquine for the prevention of malaria infection during pregnancy will be investigated in 120 women. Women will be randomized to receive either (i) 3 daily doses of AZI plus PQ, or, (ii) single dose sulfadoxine-pyrimethamine Participants will be actively followed for a period of 42 days (1, 2, 3, 4, 7, 14, 21, 28 and 42 days after treatment). At each follow-up time point the participant will have a clinical examination, fundal height measurement and assessment of foetal lie, perform a symptoms questionnaire, blood film for malaria and other scheduled safety tests (eg. Hb, glucose, ultrasound). A single blood sample for pharmacokinetic analysis will be collected at Day 4. At delivery all participants and their babies will be assessed, including blood sample for Hb, glucose, blood spot for PCR, cord blood and maternal blood. Breast milk samples will be collected for 2 weeks (Day 1, 2, 3, 4, 7, 14) after the establishment of lactation.

SECONDARY OUTCOMES:
Pharmacokinetics - distribution, terminal elimination and absorption half-life(t1/2) of azithromycin and piperaquine | 42 days intensive follow-up, final end-point at 2 weeks post delivery
Pharmacokinetics - area under the plasma concentration versus time curve (AUC) of azithromycin and piperaquine | 42 days intensive follow-up, final end-point at 2 weeks post delivery
Pharmacokinetics - peak plasma concentration (Cmax) of azithromycin and piperaquine | 42 days intensive follow-up, final end-point at 2 weeks post delivery
Pharmacokinetics - clearance (CL) of azithromycin and piperaquine | 42 days intensive follow-up, final end-point at 2 weeks post delivery
Pharmacokinetics - volume of distribution (Vd) of azithromycin and piperaquine | 42 days intensive follow-up, final end-point at 2 weeks post delivery
PCR adjusted 28 day cure | 28 days
PCR adjusted 42 day cure | 42 days
Number of participants with adverse events as a measure of safety and tolerability | 42 days intensive follow-up, final end-point at 2 weeks post delivery

OTHER OUTCOMES:
Change in maternal hemoglobin over 28 days | 28 days
Change in maternal weight over 28 days | 28 days
Infant birth weight | Time of delivery
Maternal parasitaemia | Time of delivery
Placental parasitaemia | Time of delivery
Cord blood parasitaemia | Time of delivery
Maternal hemoglobin at delivery | Time of delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Papua New Guinea Institute of Medical Research, Madang, Madang Province, Papua New Guinea